CLINICAL TRIAL: NCT07146945
Title: A Phase 1 Double-blind, Randomised, Placebo Controlled Study Evaluating the Safety, Tolerability, and Pharmacokinetics of Single Ascending Doses of S1-221 Following Oral Administration
Brief Title: A Study Testing the Safety and Effects of Single Doses of S1-221 in Healthy Volunteers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Delphian Therapeutics Australia Pty, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: DLP-S-0-1.01
Record Dates: First submitted 2025-08-02; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Healthy Participants
Keywords: Healthy Participants
MeSH Terms: interventions — Dronabinol

STUDY DESIGN:
Intervention Model Description: Part A will involve sequential ascending doses in up to 8 cohorts. Part B is a single intervention, two period, fed vs fasting comparison. Part C is an active comparator, two period crossover design. Parts B and C will only proceed after Part A has been reviewed by the Safety Review Committee (SRC) and the SRC has selected the doses for Parts B and C.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- S1-221 Single Ascending Dose (Experimental): Participants will be enrolled in 1 of 8 single ascending dose cohorts. Six participants in each cohort will receive one dose of oral S1-221.
  Doses to be administered are not pre-specified, but will be proposed, reviewed and approved by the Safety Review Committee.
  Interventions: Drug: S1-221
- Single Ascending Dose Placebo (Placebo Comparator): Two participants in each ascending dose cohort will receive one dose of oral matching placebo.
  Interventions: Drug: Placebo
- S1-221 Food Effect (Experimental): Eight participants will receive one dose of oral S1-221 under fasting conditions in Period 1 and will receive one dose of oral S1-221 under non-fasting conditions in Period 2.
  Food effect participants will be enrolled in 1 cohort. Doses to be administered are not pre-specified, but will be proposed, reviewed and approved by the Safety Review Committee.
  Interventions: Drug: S1-221
- Placebo Food Effect (Placebo Comparator): Two participants will receive one dose of oral matching placebo under fasting conditions in Period 1 and will receive one dose of oral matching placebo under non-fasting conditions in Period 2.
  Food effect participants will be enrolled in 1 cohort.
  Interventions: Drug: Placebo
- THC - active comparator crossover (Active Comparator): Five participants will receive one dose of oral THC in Period 1 and will receive one dose of oral S1-221 in Period 2.
  Participants will be enrolled in 1 cohort. The dose will be based on review of single ascending doses by the Safety Review Committee.
  Interventions: Drug: S1-221; Drug: THC
- S1-221 crossover (Experimental): Five participants will receive one dose of oral S1-221 in Period 1 and will receive one dose of oral THC in Period 2.
  Participants will be enrolled in 1 cohort. The dose will be based on review of single ascending doses by the Safety Review Committee.
  Interventions: Drug: S1-221; Drug: THC

INTERVENTIONS:
Drug: S1-221 — S1-221 will be administered orally to participants.
  Arms: S1-221 Food Effect; S1-221 Single Ascending Dose; S1-221 crossover; THC - active comparator crossover
Drug: Placebo — Matching placebo will be administered orally to participants.
  Arms: Placebo Food Effect; Single Ascending Dose Placebo
Drug: THC — A single dose of THC will be administered to participants orally.
  Arms: S1-221 crossover; THC - active comparator crossover

SUMMARY:
The purpose of this Phase 1 study is to evaluate the safety, tolerability, and pharmacokinetics (PK) profile of single ascending doses of S1-221 administered orally to healthy adult participants. S1-221 is a liquid containing cannabidiol (CBD) and Δ9-tetrahydrocannabinol (THC).

Acute subjective effects will be evaluated as a pharmacodynamic (PD) assessment and changes in plasma endocannabinoid levels will be assessed as an exploratory objective.

Data from this study will be used to select doses to be evaluated in subsequent studies to investigate the efficacy and safety of S1-221 in migraine patients.

DETAILED DESCRIPTION:
This is a first-in-human, Phase 1, randomised, double-blind study to evaluate safety, tolerability, PK, and PD following the oral administration of single ascending doses (SAD) of S1-221 to fasted and fed healthy participants.

Due to known sex differences in CBD metabolism, every effort will be made to enrol an equal number of biological females and males in each cohort (ideally no fewer than 30% females in each cohort). Individuals will only be permitted to participate in 1 study part.

Up to 10 cohorts of 8-10 participants each will be enrolled into this study. The study will consist of 3 parts. Part A will be a SAD evaluation in up to 8 cohorts. Eligible participants will be randomised in a ratio of 3:1 to receive a single oral dose of S1-221 or placebo on Day 1. Within each cohort, a sentinel group of 2 participants, randomised 1:1 to S1-221 or placebo, will be dosed at least 24 hours prior to the remaining participants in the cohort. The minimum 24-hour safety data for these sentinels will be reviewed by the Investigator, and if the dosing is deemed to be safe and well tolerated, the remaining participants in the cohort will be dosed. Study drug will be administered in a fasted state. The study duration for each fasted cohort participant will be approximately 35 days.

Parts B and C will proceed at the discretion of the Sponsor, and after review of 4 or more cohorts from Part A. Doses evaluated in Part B and C will not exceed those evaluated in Part A.

Part B will be a crossover evaluation, with and without food. Participants in Part B will be administered S1 221 or placebo once on Day 1 under fasted conditions and once on Day 15 under fed conditions. The 2 periods will be separated by a washout period of at least 14 days. A sentinel group of 2 participants, randomised 1:1 to S1-221 or placebo, will be dosed at least 24 hours prior to the remaining participants in the cohort. The minimum 24-hour safety data for these sentinels will be reviewed by the Investigator, and if the dosing is deemed to be safe and well tolerated, the remaining participants in the cohort will be dosed.

Participants in the Food Effect Cohort will be screened and administered a single oral dose of S1-221 or placebo under fasted conditions on Day 1. Participants will be discharged on Day 3 and return for an outpatient follow-up visit on Day 4 and Day 7 (+/- 2 days).

Following a washout period of at least 14 days after administration of the first dose, participants will be re-admitted 1 day prior to the second (fed) administration of study drug. On Day 15, participants will receive the same dose as in Period 1, this time following consumption of a standardised, FDA-compliant high-fat, high-calorie meal.

The study duration for each Food Effect Cohort participant will be approximately 49 days.

Part C will be a crossover evaluation of S1-221 compared to THC alone. Participants in the Part C cohort will be randomised 1:1 to treatment sequence (S1-221/THC or THC/S1-221) and administered the first treatment assignment on Day 1 and the alternative assigned drug on Day 15. The 2 periods will be separated by a washout period of at least 14 days. Both doses will be administered in a fasted state and no sentinel dosing will be performed in Part C.

The study duration for each Active Comparator Cohort participant will be approximately 49 days.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated participant informed consent form (PICF) and willing and able to follow all study procedures and requirements for the duration of the study.
* Healthy adult males and females aged 18 to 65 years, inclusive, at Screening.
* Body mass index (BMI) of 18 to 32.0 kg/m2, inclusive, and body weight ≥50.0 kg, at Screening.
* Considered healthy, as determined by no clinically significant findings from medical history or physical examination at Screening and Day -1, in the opinion of the Investigator.
* Vital signs after 5 minutes resting in supine position within the following ranges (assessment may be repeated once per schedule time point, at the discretion of the Investigator, to obtain a clinically reliable result):

  * Systolic blood pressure: 90 to 140 mmHg inclusive;
  * Diastolic blood pressure: 40 to 90 mmHg inclusive;
  * Heart rate: 40 to 100 bpm inclusive.
* Standard 12-lead ECG with parameters (average of triplicate readings) after 10 minutes in supine position within the following ranges (assessment may be repeated once per schedule time point, at the discretion of the Investigator, to obtain a clinically reliable result):

  * QRS <120 msec;
  * QT <500 msec;
  * QTc ≤450 msec (both genders);
  * PR interval ≥120 to ≤220 msec.
* Screening and Day -1 (and Day 14 for Parts B and C) safety laboratory test values within normal ranges. Out of normal range values may be accepted by the Investigator if not considered clinically significant, with the exception of the following:

  * ALT or AST >1.5 x upper limit of normal (ULN);
  * Total, indirect, or direct bilirubin >1.5 x ULN. Participants with Gilbert's syndrome with indirect bilirubin outside of the normal range will not be excluded from the study;
  * Abnormal kidney function, as assessed by estimated glomerular filtration rate (eGFR) calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI);
  * Creatinine >1.2 x ULN;
  * Haemoglobin <100.0 g/L in females or <115 g/L in males; or white blood cells <3.5 x 109/L or >11.5 x 109/L;
  * HbA1c ≥6.5% (participant must be non-diabetic). In Parts B and C, any laboratory abnormalities noted prior to the crossover repeat dosing will be discussed with the medical monitor and Sponsor to determine whether repeat dosing may proceed as planned.
* Negative tests for HBsAg, HBcAb, anti-HCV, and HIV antibodies at Screening.
* Women of childbearing potential (WOCBP) must have a negative pregnancy test at Screening and Day -1 (and Day 14 for Parts B and C).

Note: Definition of child-bearing potential is fertile and following menarche until becoming post-menopausal, unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A post-menopausal state is defined as no menses for 12 months without an alternative medical cause and follicle-stimulating hormone (FSH) documented in the post- menopausal range (≥40 IU/L).

* WOCBP must agree to the use adequate contraception from Screening through 60 days following the last dose of study drug. Additionally, they should avoid egg/ova donation throughout the study and for 60 days after the last dose of the study drug.
* Male participants must agree to use adequate contraception from Screening through 95 days following the last dose of study drug. Male participants with female partners that are surgically sterile or post-menopausal (defined as being amenorrhoeic for at least 12 months without an alternative medical cause) may also be included and will not be required to use above-described methods of contraception. Male partners with potentially post-menopausal females who are under the age of 55 years must use condoms unless their partner's postmenopausal status has been confirmed by FSH level >40mIU/mL. Male participants who have undergone vasectomy and have had testing to confirm azoospermia 90 days after procedure may also be included. The use of condom by male participant will be required if vasectomy is the chosen highly effective method of contraception. Male participants must also agree not to donate sperm throughout the study and for 95 days following the last dose of study drug.
* Non-smoker, ex-smoker, or smoker willing to refrain from use of tobacco/nicotine-containing products, e.g., cigarettes, vaporizers, cigars, pipe tobacco, smokeless tobacco, nicotine gum, lozenges, patches, on more than 5 occasions within 1 month prior to the Screening visit and for the duration of the study. Note: a cotinine level or other observations that, in the opinion of the Investigator, suggest heavy use of tobacco will be exclusionary.
* Willing to refrain from consumption of alcohol as follows:

  * Part A: for at least 48 hours prior to Screening and Day -1, then from Day 1 through End of Study (EOS).
  * Parts B and C: for at least 48 hours prior to Screening, Day -1, and Day 14, and from Day -1 through Day 7 visit, and from Day 14 through EOS (consumption of alcohol is permitted from Day 8 through Day 13).
* Willing to withhold cannabinoids (including CBD and THC) and cannabis (including hemp) products for 60 days prior to administration of the first dose of study drug and throughout the study.
* Willing to refrain from consumption of food or beverages containing xanthine derivatives or xanthine-related compounds (e.g., coffee, black/green tea, chocolate) or energy drinks from 48 hours prior to each clinic admission and each follow-up visit.
* Willing to defer blood donations to a blood service for minimum of 30 days following the last dose of study drug.
* Willing to comply with the study-specified diet while confined in the CRU. Participants in Part B (Food Effect Cohort) must agree to complete consumption of a standardised high-fat, high-calorie breakfast during the fed period on Day 15.
* Willing to not operate a motor vehicle or heavy machinery for 7 days following administration of study drug.
* In the opinion of the Investigator, is willing and able to comply with and understand study requirements and be available for the required study visits.

Exclusion Criteria:

* Female participant who is pregnant or breastfeeding, or planning to become pregnant or breastfeed during study participation.
* Evidence of clinically significant abnormalities or disease, including, but not limited to, the following:

  * Any pulmonary, cardiovascular, neurologic, gastrointestinal, hepatic, renal, endocrine or other disease, at the discretion of the Investigator including, but not limited to, history of epilepsy.
  * Any history of gastrointestinal condition, including surgeries, or use of any medications (including glucagon-like peptide-1 [GLP-1] agonists) which may affect absorption or gastric motility after oral administration.
  * Has a lifetime history or current diagnosis of a significant psychiatric disorder including, but not limited to, schizophrenia spectrum or other psychotic disorders, major depressive disorder, or generalized anxiety disorder per Diagnostic and Statistical Manual of Mental Disorders 5th Edition (DSM-5), and/or has first-degree relative with a history of psychosis or schizophrenia.
  * Meets DSM-5 criteria for lifetime or current substance use disorder for any psychoactive substances other than nicotine or caffeine.
  * Has a history of, or active, suicidal ideation as identified by positive response to questions 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) at Screening, or has any prior history of suicidal behaviour, as evidenced by medical history of suicide attempt or a "Yes" response to the following suicidal behaviour questions on the C-SSRS: actual attempt, interrupted attempt, or aborted attempt.
  * History or ECG evidence of myocardial ischemia or infarct, 2nd or 3rd degree AV block, bundle branch block, with the exception of incomplete right bundle branch block in the absence of clinical heart disease, or multiple or multifocal premature ventricular contractions.
  * History of fainting or syncope that, in the Investigator's opinion, would interfere with study conduct or compliance.
  * Any other laboratory, vital sign, ECG abnormality, or clinical history or finding that, in the Investigator's opinion, is likely to unfavourably alter the risk-benefit of study participation, confound study results, or interfere with study conduct or compliance.
* Positive urine drug test or alcohol breath test at Screening or Day -1 (and Day 14 for the Parts B and C), unless there is an explanation deemed acceptable by the Investigator and/or the participant tests negative upon re-test. Note: one re-test for drug screen is permitted per scheduled time point. No retest is permitted for alcohol breath test.
* History of clinically significant allergy, hypersensitivity, or adverse reaction to cannabis or any cannabinoid, including dysphoria, or to any excipient in the investigational product (e.g., sesame allergy) at the discretion of the Investigator.
* Donation or loss of greater than 1 unit (450 mL) of blood within the 4 weeks prior to Screening.
* Has received any prescription medication within 14 days or 5 half-lives (whichever is longer) of Day -1 and throughout the study (exceptions: contraceptives are permitted). Prescriptions of known inhibitors or inducers of hepatic drug metabolism (e.g., rifampin, carbamazepine, phenytoin, barbiturates [e.g., phenobarbital and butalbital], dexamethasone, antidepressants [e.g., fluoxetine, paroxetine], proton pump inhibitors, ketoconazole itraconazole and clarithromycin) will be prohibited.
* Has received any non-prescription medication within 5 days of Day -1 and throughout the study (exception: occasional [PRN] paracetamol [up to 2 g/day] or ibuprofen [up to 1.2 g/day] use may be permitted, at Investigator discretion).
* Use of vitamins, natural and herbal remedies including St. John's wort, supplements (including kratom), or vaccines in the 14 days prior to Day -1 and throughout the study.
* Use of any investigational drug within 30 days or <5 half-lives, whichever is longer, prior to administration of first dose of study drug and throughout the study.
* Consumption of grapefruit, starfruit, pomegranate, pomelo, pineapple, or Seville orange, products in the 7 days prior to Day -1 until completion of the EOS visit.
* Regular alcohol consumption in excess of 14 units per week or 2 standard drinks in a single day. One standard drink is defined as containing 10 grams of pure alcohol, e.g., 285 mL normal-strength beer (4.9% alcohol), 100 mL of non-fortified wine (13% alcohol), or 30 mL of spirits (40% alcohol).
* Behaviour suggestive of unreliability or inability to comply with study requirements per discretion of the Investigator.
* Identified as a site employee of the Investigator or study centre, with direct involvement in the proposed study or other studies under the direction of that Investigator or study centre, as well as family members (i.e., immediate, husband, wife or de facto and their children, adopted or natural) of the site employees or the Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2026-02-22 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with treatment-emergent Adverse Events (AE). An AE will be considered treatment-emergent if the onset date and time is at the time of or after first study drug administration. | Through to study completion, up to approximately 49 days.
  Incidence, severity and relationship of AEs.
Percentage of participants with treatment-emergent abuse-related Adverse Events (AE). An AE will be considered treatment-emergent if the onset date and time is at the time of or after first study drug administration. | Through to study completion, up to approximately 49 days.
  Incidence, severity and relationship of abuse-related AEs.
Percentage of participants with out-of-range red blood cell count (cells/µL). | Through to study completion, up to approximately 49 days.
  Changes from baseline in red blood cell count (cells/µL).
Percentage of participants with out-of-range haematocrit (L/L). | Through to study completion, up to approximately 49 days.
  Changes from baseline in haematocrit (L/L).
Percentage of participants with out-of-range haemoglobin (g/L). | Through to study completion, up to approximately 49 days.
  Changes from baseline in haemoglobin (g/L).
Percentage of participants with out-of-range white blood cell count including differential count (neutrophils, eosinophils, basophils, monocytes, and lymphocytes) (cells/µL). | Through to study completion, up to approximately 49 days.
  Changes from baseline in white blood cell count including differential count (neutrophils, eosinophils, basophils, monocytes, and lymphocytes) (cells/µL).
Percentage of participants with out-of-range platelets (cells/µL). | Through to study completion, up to approximately 49 days.
  Changes from baseline in platelets (cells/µL).
Percentage of participants with changes from baseline in Sodium (mmol/L). | Through to study completion, up to approximately 49 days.
  Changes from baseline in Sodium (mmol/L).
Percentage of participants with changes from baseline in Potassium (mmol/L). | Through to study completion, up to approximately 49 days.
  Changes from baseline in Potassium (mmol/L).
Percentage of participants with changes from baseline in Chloride (mmol/L). | Through to study completion, up to approximately 49 days.
  Changes from baseline in Chloride (mmol/L).
Percentage of participants with changes from baseline in Calcium (mmol/L). | Through to study completion, up to approximately 49 days.
  Changes from baseline in Calcium (mmol/L).
Percentage of participants with changes from baseline in Bicarbonate (mmol/L). | Through to study completion, up to approximately 49 days.
  Changes from baseline in Bicarbonate (mmol/L).
Percentage of participants with changes from baseline in Magnesium (mmol/L). | Through to study completion, up to approximately 49 days.
  Changes from baseline in Magnesium (mmol/L).
Percentage of participants with changes from baseline in Aspartate transaminase (U/L). | Through to study completion, up to approximately 49 days.
  Changes from baseline in Aspartate transaminase (U/L).
Percentage of participants with changes from baseline in Alanine Transaminase (U/L). | Through to study completion, up to approximately 49 days.
  Changes from baseline in Alanine Transaminase (U/L).
Percentage of participants with changes from baseline in Alkaline Phosphatase (U/L). | Through to study completion, up to approximately 49 days.
  Changes from baseline in Alkaline Phosphatase (U/L).
Percentage of participants with changes from baseline in Gamma-Glutamyl Transferase (U/L). | Through to study completion, up to approximately 49 days.
  Changes from baseline in Gamma-Glutamyl Transferase (U/L).
Percentage of participants with changes from baseline in Lactate dehydrogenase(U/L). | Through to study completion, up to approximately 49 days.
  Changes from baseline in Lactate dehydrogenase(U/L).
Percentage of participants with changes from baseline in Bilirubin (µmol/L). | Through to study completion, up to approximately 49 days.
  Changes from baseline in Bilirubin (µmol/L).
Percentage of participants with changes from baseline in urea (mmol/L). | Through to study completion, up to approximately 49 days.
  Changes from baseline in urea (mmol/L).
Percentage of participants with changes from baseline in Creatinine (µmol/L). | Through to study completion, up to approximately 49 days.
  Changes from baseline in Creatinine (µmol/L).
Percentage of participants with changes from baseline in Phosphorus (mmol/L). | Through to study completion, up to approximately 49 days.
  Changes from baseline in Phosphorus (mmol/L).
Percentage of participants with changes from baseline in Uric acid (mmol/L). | Through to study completion, up to approximately 49 days.
  Changes from baseline in Uric acid (mmol/L).
Percentage of participants with changes from baseline in glucose (mmol/L). | Through to study completion, up to approximately 49 days.
  Changes from baseline in glucose (mmol/L).
Percentage of participants with changes from baseline in HbA1c (%). | Through to study completion, up to approximately 49 days.
  Changes from baseline in HbA1c (%).
Percentage of participants with changes from baseline in Albumin (g/L). | Through to study completion, up to approximately 49 days.
  Changes from baseline in Albumin (g/L).
Percentage of participants with changes from baseline in Total protein (g/L). | Through to study completion, up to approximately 49 days.
  Changes from baseline in Total protein (g/L).
Percentage of participants with changes from baseline in Globulin (g/L). | Through to study completion, up to approximately 49 days.
  Changes from baseline in Globulin (g/L).
Percentage of participants with changes from baseline in Cholesterol (mmol/L). | Through to study completion, up to approximately 49 days.
  Changes from baseline in Cholesterol (mmol/L).
Percentage of participants with changes from baseline in Triglycerides (mmol/L). | Through to study completion, up to approximately 49 days.
  Changes from baseline in Triglycerides (mmol/L).
Percentage of participants with changes from baseline in Creatine Kinase (U/L). | Through to study completion, up to approximately 49 days.
  Changes from baseline in Creatine Kinase (U/L).
Percentage of participants with changes from baseline in C-reactive protein (mg/L). | Through to study completion, up to approximately 49 days.
  Changes from baseline in C-reactive protein (mg/L).
Percentage of participants with changes from baseline in Estimated Glomerular Filtration Rate (mL/min/1.73m2). | Through to study completion, up to approximately 49 days.
  Changes from baseline in Estimated Glomerular Filtration Rate (mL/min/1.73m2).
Percentage of participants with changes from baseline in Thyroid Stimulating Hormone (mIU/L). | Through to study completion, up to approximately 49 days.
  Changes from baseline in Thyroid Stimulating Hormone (mIU/L).
Percentage of participants with changes from baseline in Activated Partial Thromboplastin Time (sec). | Through to study completion, up to approximately 49 days.
  Changes from baseline in Activated Partial Thromboplastin Time (sec).
Percentage of participants with changes from baseline in Prothrombin Time (sec). | Through to study completion, up to approximately 49days.
  Changes from baseline in Prothrombin Time (sec).
Percentage of participants with changes from baseline in International Normalised Ratio (ratio). | Through to study completion, up to approximately 49days.
  Changes from baseline in International Normalised Ratio (ratio).
Percentage of participants with changes from baseline in urinalysis laboratory parameters. Assessment from the patient through dipstick testing on a freshly voided urine sample to measure the presence or absence of protein glucose, blood (erythrocytes), | Through to study completion, up to approximately 49days.
  Changes from baseline in urinalysis laboratory parameters. Assessment from the patient through dipstick testing on a freshly voided urine sample to measure the presence or absence of protein glucose, blood (erythrocytes), leucocytes, ketone bodies, nitrite, bilirubin, urobilinogen (present/absent).
Percentage of participants with changes from baseline in urine pH. | Through to study completion, up to approximately 49days.
  Changes from baseline in urine pH.
Percentage of participants with changes from baseline of systolic and diastolic blood pressure, measured in mmHg. | Through to study completion, up to approximately 49days.
  Changes from baseline of systolic and diastolic blood pressure, measured in mmHg.
Percentage of participants with changes from baseline heart rate, measured in beats per minute (bpm). | Through to study completion, up to approximately 49days.
  Changes from baseline heart rate, measured in beats per minute (bpm).
Percentage of participants with changes from baseline respiratory rate, measured in breaths per minute. | Through to study completion, up to approximately 49days.
  Changes from baseline respiratory rate, measured in breaths per minute.
Percentage of participants with changes from baseline body temperature, measured in degrees Celsius. | Through to study completion, up to approximately 49days.
  Changes from baseline body temperature, measured in degrees Celsius.
Percentage of participants with changes from baseline of 12-lead ECG parameters. The following parameters are included: heart rate, RR interval, PR interval, QRS duration, QT interval, and QTcF interval (all measured in mV/s). | Through to study completion, up to approximately 49days.
  Changes from baseline of 12-lead ECG parameters. The following parameters are included: heart rate, RR interval, PR interval, QRS duration, QT interval, and QTcF interval (all measured in mV/s).
Percentage of participants with changes from baseline in physical examination measured by presence or absence of investigator-assessed abnormalities. | Through to study completion, up to approximately 49days.
  Changes from baseline in physical examination measured by presence or absence of investigator-assessed abnormalities. The following parameters are included: general appearance, head, ears, eyes, nose, throat, dentition, thyroid, chest (heart, lungs), abdomen, skin/soft tissues, neurological, extremities, back, neck, musculoskeletal, and lymph nodes.
Percentage of participants with changes from baseline in suicidal ideation and behaviour as assessed by Columbia-Suicide Severity Rating Scale with scoring is based on the most severe response reported for suicidal ideation and behaviours. | Through to study completion, up to approximately 49 days.
  Changes from baseline in suicidal ideation and behavior as assessed by Columbia-Suicide Severity Rating Scale with scoring is based on the most severe response reported for suicidal ideation and behaviours. Suicidal ideation will be reported with scores of 0-25, with 0 being no suicidal ideation and 25 being the most severe ideation. Behaviour will be reported in terms of presence or absence, frequency, and their severity (actual attempt, interrupted/aborted attempt, or mere preparation).

SECONDARY OUTCOMES:
Pharmacokinetics parameter - maximum observed concentration (Cmax) | Through to study completion, up to approximately 49 days.
  Maximum observed plasma concentration (Cmax) of S1-221 and its metabolites.
Pharmacokinetics parameter - Time for maximum observed Concentration (Tmax). | Through to study completion, up to approximately 49 days.
  Time to maximum observed plasma concentration (Tmax) of S1-221 and its metabolites.
Pharmacokinetics parameter - Area under the curve (AUC) | Through to study completion, up to approximately 49 days.
  Area under the plasma concentration-time curve (AUC) of S1-221 and its metabolites from time 0 (time of dosing) to time of the last quantifiable concentration
Pharmacokinetics parameter - Elimination rate constant | Through to study completion, up to approximately 49 days.
  Elimination rate constant (Kel) of S1-221 and its metabolites. The elimination rate constant is a value used in pharmacokinetics to describe the rate at which a drug is removed from the system.
Pharmacokinetics parameter - Apparent total plasma clearance | Through to study completion, up to approximately 49 days.
  Apparent total plasma clearance (CL/F) of S1-221 and its metabolites.
Pharmacokinetics parameter - Apparent volume of distribution | Through to study completion, up to approximately 49 days.
  Apparent volume of distribution (Vx/F) of S1-221 and its metabolites.
Pharmacokinetics parameter - dose corrected maximum observed concentration | Through to study completion, up to approximately 49 days.
  Dose-corrected maximum observed plasma concentration (Cmax/Dose) of S1-221 and its metabolites.
Pharmacokinetics parameter - dose corrected area under the plasma concentration-time curve | Through to study completion, up to approximately 49 days.
  The dose-corrected area under the plasma concentration-time curve (AUC/Dose) of S1-221 and its metabolites.
Pharmacokinetics - cumulative amount of S1-221 excreted unchanged in urine | Through to Day 3.
  The cumulative amount of S1-221 excreted unchanged in urine will be measured for all participants.
Pharmacokinetics - fraction of S1-221 dose excreted unchanged into urine as a percentage | Through to Day 3.
  The fraction of S1-221 dose excreted unchanged into urine (Fe%) will be measured for all participants, as a percentage.
Pharmacokinetics - renal clearance of S1-221 | Through to Day 3.
  The renal clearance of S1-221 (CLr) will be measured for all participants.
Pharmacodynamic (PD) effects | Up to 12 hours post administration of S1-221.
  Subjective drug effects following single oral doses of S1-221 will be assessed by asking participants, "Do you feel a drug effect right now," rated using a unipolar 100 mm visual analogue scale, with anchors of "not at all" on one end and "extremely" on the other.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Lanier, Study Chair — DelphianTherapeutics
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No